The Statistical Package for Social Sciences (SPSS) for Windows 20 was used for statistical analysis (IBM SPSS Inc., Chicago, IL). The Kolmogorov-Smirnov test was used to determine the data's normal distribution. Numerical variables with normal distributions are represented by mean±standard deviation, while numerical variables with non-normal distributions are represented by median (min-max). Numbers and percentages are used to represent categorical variables. The Student's T test was used for parametric values and the Mann-Whitney U test was used for nonparametric values when comparing numerical variables between the two groups. To compare categorical variables, the Chi-square test was used. The changes in numerical variables in the postoperative follow-up, as well as the differences in these changes between the control and experimental groups, were examined using mixed model analysis in repeated measurements. Cochran's Q test was used to examine changes in categorical variables (post hoc test: McNemar test). In statistical analysis, the p=0.05 value was accepted as significant.